CLINICAL TRIAL: NCT05763186
Title: The Right Amount of Purge Useful for Blood Sampling on PiccLine
Brief Title: The Right Amount of Purge Useful for Blood Sampling on PiccLine (PiccLine)
Acronym: PiccLine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC22_9907-2_PiccLine; 2022-A01383-40 (Other: N°ID-RCB)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-09

CONDITIONS: Hematology
Keywords: PiccLine; blood collection; purge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sampling (Experimental): * On the PiccLine: a collection of 6 consecutive heparinized tubes with 3.5ml gel corresponding to the usual purge volume
  * In the periphery : one 3.5ml heparin-gel tube as a reference.
  Interventions: Other: Sampling
- Sampling and rinsing (Experimental): * On the PiccLine: a 10 ml pre-rinsing with 0.9% NaCl and then a sampling of 6 consecutive heparinized tubes with 3.5ml gel corresponding to the usual purge volume.
  * In the periphery: one 3.5 ml heparin-gel tube as a reference.
  Interventions: Other: Sampling and rinsing

INTERVENTIONS:
Other: Sampling — Comparison of the results of the biological examinations obtained on the 6 tubes collected on the PiccLine with the results of the biological examinations obtained on the peripheral sample.
  Arms: Sampling
Other: Sampling and rinsing — Comparison of the results of the biological examinations obtained on the 6 tubes collected on the PiccLine with the results of the biological examinations obtained on the peripheral sample.
  Arms: Sampling and rinsing

SUMMARY:
An increasing number of patients are receiving central lines, including PiccLine systems for the administration of therapeutics and nutrition.

Although these systems are not theoretically intended for blood collection, nurses prefer them as a puncture site when they are in place in their patients, saving them from further peripheral puncture in people who generally do not have optimal venous capital.

It is essential to purge the tubing in place in the patient and filled with infusion solution before drawing blood. Although the dead volume of the tubing used does not exceed 2mL, the volume of purging required before filling tubes for the laboratory appears to be much greater. Anecdotal evidence suggests a useful volume of 20ml but this has never been clearly demonstrated. In addition, the Biochemistry laboratory regularly sees blood samples diluted with perfusion solution, as evidenced by biochemical assays, leading to the cancellation of analyses received in the laboratory and a new sample being taken. This increases blood spoliation for these often already anaemic patients.

There is no consensus in the literature on recommendations for such sampling in PiccLine patients:

* The CLSI1 (Clinical and Laboratory Standart Institute), a non-governmental organisation, issued sampling recommendations in 2017 that were taken up by Becton Dickinson2, a supplier of blood collection tubes. These recommendations include:

  * Rinse with 10 ml of 0.9% NaCl
  * Then a purge of 3 to 11 ml (depending on the analysis sought)
* English-language articles3,4,5,6,7 show purge volumes ranging from 3 to 6 ml with significantly different sampling methods (rinsing or not).

The investigators therefore note a discrepancy between the sampling practices of the university hospital and the recommendations of the CLSI. In fact, the investigators noted a lack of rinsing prior to purging, which could explain the difference between 20 and 3 ml. This raises the issue of protocolisation of this type of sampling in order to standardise practices.

A consultation of other hospitals, carried out beforehand, enabled us to note that French practices are not in agreement with these recommendations. The management of the Rennes University Hospital as well as the Haute Autorité de Santé were contacted in order to confirm that no normative document had been published or was being drafted on this subject.

The fields of study are: sampling practices on PiccLine, the pre-analytical phase in medical biology.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Carrier of PiccLine one way polyurethane
3. Hospitalized in a clinical hematology unit This criterion minimises patient and practice heterogeneity.
4. PiccLine placement not older than 48 hours
5. Injection of at least one solution
6. Affiliated to a social security scheme
7. Having signed a free, informed and written consent

Exclusion Criteria:

1. Anemia below the transfusion threshold (hemoglobin level < 7 g/dL) in relation to the patient's pathology
2. Parenteral nutrition
3. Peripheral venous sampling not possible (insufficient venous capital)
4. Protected person (adult subject to legal protection (safeguard of justice, curatorship, guardianship), person deprived of liberty, pregnant woman (declarative), breastfeeding woman and minor).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Lowest purge volume to obtain a biological result in the PiccLine sample that matches the peripheral sample taken from the same patient at the same time for the following assays: - Sodium, potassium and chlorine - Creatinine - Glucose | during 2 days follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eric Geffray, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France